CLINICAL TRIAL: NCT03538886
Title: The Nordic-Baltic Heart Team Initiative for Improved Long-term Coronary Artery Revascularization Outcome in Patients With Proximal Left Descending Coronary Artery (LAD) Lesion. NOBLE LAD
Brief Title: Nordic-Baltic Coronary Revascularization Study in Patients With Proximal Left Descending Coronary Artery (LAD) Lesion.
Acronym: NOBLE-LAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossible to involve a sufficient number of centers in the study.
Sponsor: Aalborg University Hospital (Other)
Collaborators: Oulu University Hospital (Other); Region Örebro County (Other); Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Principal Investigator, Leif Thuesen, Senior interventional cardiologist, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOBLE-LAD_Protocol version 3
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary revascularization
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: 1:1 randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The clinical outcomes will be assessed by an independent event committee with no knowledge of treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous coronary intervention (PCI) (Active Comparator): Currently, percutaneous coronary intervention (PCI) using balloon and drug eluting stents is the treatment of choice for treatment of a proximal LAD lesion.
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- Coronary artery bypass grafting (CABG) (Experimental): Coronary artery bypass grafting is a well established treatment with documented excellent long-term results for the treatment of proximal LAD lesion.
  Interventions: Procedure: Coronary artery bypass grafting (CABG)

INTERVENTIONS:
Procedure: Coronary artery bypass grafting (CABG) — Revascularization of LAD lesion by CABG
  Arms: Coronary artery bypass grafting (CABG)
Procedure: Percutaneous coronary intervention (PCI) — Revascularization of LAD lesion by PCI
  Arms: Percutaneous coronary intervention (PCI)

SUMMARY:
The Nordic-Baltic Heart Team Initiative for improved long-term coronary artery revascularization outcome compares quality of life and survival after coronary bypass grafting (CABG) vs. percutaneous coronary intervention (PCI) in patients with 1-vessel disease and proximal stenosis of the anterior descending artery (LAD/in patients with isolated proximal left descending coronary artery (LAD) lesion

DETAILED DESCRIPTION:
It is not clear how operable 1-VD patients with stable or stabilized coronary artery disease involving a pLAD lesion should be treated to optimize long-term survival and quality of life.

According to recent European guidelines, significant pLAD disease may be treated by PCI or by CABG. This recommendation is based on two meta-analyses including 1.210 and 1.952 randomized and non-randomized patients. Generally, the patients were followed for 4-5 years. The analyses reported similar rates of mortality, MI and stroke, but more repeat revascularizations after PCI. Only one study including129 patients provided more than 5-year follow-up. Thus, the there is limited documentation for long-term effect of PCI vs. surgical re-vascularization in pLAD disease.

The American 2014 Guidelines on coronary revascularization recommends CABG for improved survival in patients with solitary proximal LAD stenosis. CABG

The angiographic 90% LIMA patency rate after 1, 2 and 3 decades is well described and suggestive of a survival benefit of surgical revascularization.

Therefore, there is scientific background for an CABG LIMA-to-LAD vs. PCI comparison in 1-VD patients with a pLAD lesion.

Substantiated expectations:

* PCI is superior to bypass operation concerning short-term quality of life.
* Off-pump LIMA-to-LAD is superior to PCI concerning long-term all-cause mortality.
* Long-term (≥10-year) follow-up is essential to evaluate coronary revascularization strategies.
* Outcome may be dependent on lesion complexity, diabetes and gender.

ELIGIBILITY:
Inclusion Criteria:

Heart Team decision on treatment

1-VD patients with stable coronary artery disease or stabilized unstable angina pectoris/NSTEMI or silent ischemia Proximal LAD (pLAD) stenosis (>90% by visual assessment or FFR <80% The lesion may be treated by both PCI and surgery

Exclusion Criteria:

ST-elevation myocardial infarction within 24 hours. Expected survival <1 year, because of high age or severe cardiac or non-cardiac disease.

Significant LM disease. Earlier CABG. PCI within 3 months. Significant valvular heart disease. Renal failure on dialysis Earlier disabling stroke Relative or absolute contraindication to dual antiplatelet therapy. Allergy relevant to the study treatments. Age < 18 years. Study required information and consent suboptimal or impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 10 years
  Death of any cause
Quality of life | 1 year
  By SF 12 and Seatle Angina Questionaire
MACCE | 1 year
  Major cardiac and cerebral adverse events (myocardial infarction, stroke, revascularization, death)

SECONDARY OUTCOMES:
All-cause death | 1, 2, 3, 5 and 10 years
  Death of any cause
Cardiac death | 1, 2, 3, 5 and 10 years
  Death of cardiac disease
Spontaneous myocardial infarction | 1, 2, 3, 5 and 10 years
  Type 1 myocardial infarction
Procedure related myocardial infarction | 1, 2, 3, 5 and 10 years
  Myocardial infarction related to PCI or CABG
Major stroke, minor stroke and al stroke | 1, 2, 3, 5 and 10 years
  Stroke by VARC definition
Angina | 1, 2, 3, 5 and 10 years
  CCS angina class
Heart failure | 1, 2, 3, 5 and 10 years
  NYHA class
Stent thrombosis | 1, 2, 3, 5 and 10 years
  ARC-define stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Leif Thuesen, MD, Principal Investigator — Department of Cardiology, Aalborg University Hospital; Jan Jesper Andreasen, Prof, Principal Investigator — Department of Cardiothoracic Surgery, Aalborg University Hospital; Peter Sogaard, Prof, Study Chair — Department of Cardiology, aaalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After publication of the trial, data will be made available for metaanalyses on request, and after accept by the steering committee.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and statistical analysis plan available by now.
Access Criteria: At clinicaltrial.gov